CLINICAL TRIAL: NCT01117519
Title: Impact of a Balanced Infusion Solution Compound of 50% Crystalloid and 50% Colloid Versus an Unbalanced Infusion Solution of 100% Crystalloid Within a Goal-directed Hemodynamic Protocol on Acid-base Balance
Brief Title: Impact of Fluid Management Within a Goal-directed Hemodynamic Protocol on Acid-base Balance in Elective Trauma Surgery
Acronym: HIPSTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Prof. MD, Director of the Dept. of Anaesthesiology and Intensive Care Medicine, CVK, CCM, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIPSTER
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Hemodynamic Instability
Keywords: fluid and volume management; acid-base balance; goal-directed therapy; transoesophageal doppler
MeSH Terms: interventions — Home Infusion Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- unbalanced infusion solution (Active Comparator)
  Interventions: Drug: Infusion Therapy
- balanced infusion solution compound (Active Comparator)
  Interventions: Drug: Infusion Therapy

INTERVENTIONS:
Drug: Infusion Therapy — Based on changes of stroke volume measured by transoesophageal doppler patients during elective hip surgery will achieve either a unbalanced infusion solution, maximum dose of 100 ml/kg BW, or a compound of balanced infusion solution including 50% crystalloid and 50% colloid, each: maximum dose of 50 ml/kg BW. The study medication will be administered only during surgery.

SUMMARY:
The purpose of this study is to determine whether the administration of a compound of balanced infusion solutions including 50% crystalloid and 50% colloid has a positive impact on acid-base balance in elective hip replacement surgery. The application of the study medication will be carried out through a goal-directed intraoperative therapy by transoesophageal doppler.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the age of 60 and above who want to undergo an elective hip replacement surgery in the center of musculoskeletal surgery
* Offered patient information and written informed consent

Exclusion Criteria:

* Participation in another trial according to the German Drug Law 30 days to and during the study
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* (Unclear) history of alcohol or substances disabuse
* Absent knowledge of german language
* Analphabetism
* Allergy to hydroxyethyl starch or other ingredients of the intravenous solutions
* For women: Pregnancy or positive pregnancy test within the preoperative screening
* Operation due to case of emergency, polytrauma or pathologic fracture
* Only use of regional anaesthesia
* American Society of Anaesthesiologists (ASA) classification greater than III
* Peripheral or central edema
* AIDS (according to the CDC-classification of HIV-infection: category C)
* Rheumatoid disease under treatment with Anti-TNF-alpha-Ab and/or high-dose-corticoid-treatment
* Immunosuppression therapy
* History of bleeding tendency (e.g. von-Willebrand-disease, thrombocytopenia)
* Derailed metabolic disorder (e.g. Diabetes mellitus (Glucose > 300 mg/dl) during the preoperative screening)
* Known history of electrolyte disturbance (e.g. Hyperkalemia > 5.8 mmol/l, Hypernatraemia > 155 mmol/l)
* Known history of acid-base-dysbalances
* History of intracranial hemorrhage within one year of participation in the study
* Neurological or psychiatric disease with limited contractual capability
* Advanced disease of the oesophagus or upper respiratory tract
* Operation in the area of the oesophagus or nasopharynx within the last two months
* CHF (congestive heart failure) according to (New York Heart Association) classification - NYHA class IV
* Liver disease (CHILD B or C cirrhosis, end-stage liver disease (MELD-score greater than 10))
* Conditions after acute or chronic pancreatitis
* Renal insufficiency (serum creatinine greater than 2.0 mg/dl or greater than 150 µmol/l or dependency of haemodialysis)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Standard Base Excess | up to 2 days
  After administration of 2 litres of study medication. In recovery room. On general ward.

SECONDARY OUTCOMES:
SID (strong ion difference) | up to 2 days
  Change of the SID (strong ion difference) according to the stewart-approach of evalutation acid-base-dysbalances
Hemodynamic Stability | up to 6 days
  Doses and duration of therapy with catecholamins, number and duration of hypotensive episodes
Fluid Loss of Drainage | up to 6 days
  The quantity of fluids per day losing by drainage during the first three days after surgery
Discharge Criteria, Length of Hospital Stay | 5 days up to hospital discharge
  Time until fullfilling the hospital discharge criteria (measured by the postanesthesia discharge scoring system (PADSS)), and length of hospital stay
Organ Function/Dysfunction | up to 6 days
  (Cumulative) frequency of postoperative organ dysfunctions (cerebral, cardiac, pulmonary, renal, gastrointestinal)
Incidence of Infections | up to 5 days
  Perioperative Incidence of infections (according to the Centers of Disease and Prevention (CDC))
Pain | up to 6 days
  Pain of the patient measured by NAS (Numeric analogue scale), VAS (Visual analogue scale), NRS (Numeric rating scale) and BPS (Behavioral pain scale)
Incidence of Delirium | up to 6 days
  Incidence of delirium measured accordingly by DSM IV (Diagnostic and statistical manual of mental disorders criteria for delirium), Nu-DESC (Nursing delirium screening scale), DDS (Delirium detection score), CAM (Confusion assessment method), CAM-ICU (Confusion assessment method for the ICU), DRS (Delirium rating scale) and ICDSC (Intensive care delirium screening checklist).
Incidence of Postoperative Cognitive Deficit (POCD) | up to 90 days after surgery
  Measurement of cognitive function by 5 tests out of CANTAB (Cambridge neuropsychological test automated battery) modeled by the ISPOCD1 study (International study of post-operative cognitive dysfunction), Stroop colour word test(SCWT) and verbal learning test(VLT)
Mobilisation | up to 6 days
  Duration and type of mobilisation

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, Prof., MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine, Campus Charité Mitte, Charitéplatz 1, Berlin, Germany